CLINICAL TRIAL: NCT01712854
Title: Investigating the Effects of Symbicort on the Ventilatory Kinematics in Patients With Obstructive Disease With Optoelectronic Plethysmography
Brief Title: Effects of Symbicort on the Ventilatory Kinematics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closed by study sponsor; PI left the institution; responsible party changed to Columbia
Sponsor: Columbia University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAI1932
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD; Chronic Obstructive Lung Disease; Long acting beta agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort (Experimental): A combination of budesonide + long acting beta agonist (Symbicort): Budesonide 80 mcg and formoterol fumarate dihydrate inhaler 4.5 mcg
  Interventions: Drug: Symbicort
- Budesonide only (Placebo Comparator): Budesonide 80 mcg (Entocort EC) only
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — budesonide 80 mcg
  Arms: Budesonide only
Drug: Symbicort — A combination of budesonide and long acting beta agonist: Budesonide 80 mcg and formoterol fumarate dihydrate inhaler 4.5 mcg
  Arms: Symbicort

SUMMARY:
The purpose of this study is to investigate how budesonide/formoterol fumarate dihydrate (Symbicort ©) affects dynamic hyperinflation in patients with obstructive disease using Optoelectronic Plethysmography (OEP). This study is unique as it will be the first randomized, doubleblind, crossover study with a placebo inhaler and budesonide/formoterol fumarate dihydrate as the intervention which will evaluate the effects on ventilatory mechanics through the use of OEP. The investigators plan to demonstrate that budesonide/formoterol fumarate dihydrate impacts dynamic hyperinflation which can be detected with OEP, and that budesonide/formoterol fumarate dihydrate may have an effect in the short term on exercise capacity during a constant load exercise test. The changes in ventilatory mechanics measured after budesonide/formoterol fumarate dihydrate by OEP will provide a unique evaluation of budesonide/formoterol fumarate dihydrate in a controlled setting also demonstrating the utility of OEP in evaluating of the effects of a medical treatment on hyperinflation in individuals with chronic obstructive lung disease (COPD).

1. Primary Objective/Hypothesis: Our objective is to measure baseline, post treatment and post exercise spirometry and evaluate exercise dynamic hyperinflation before and after treatment using OEP. The investigators hypothesize that budesonide/formoterol fumarate dihydrate will decrease dynamic hyperinflation as measured by OEP.
2. Primary Endpoint: Our primary endpoint is the change in dynamic hyperinflation, specifically end expiratory volumes, dynamic lung volumes and diaphragmatic paradoxical breathing as measured by OEP.
3. Secondary Objective: Our secondary objective is to evaluate duration of steady state exercise and exercise capacity before and after treatment. Our secondary hypothesis is that decreases in dynamic hyperinflation during exercise will lead to improvements in dyspnea with exercise, and allow for increases in exercise capacity.
4. Secondary endpoint: Exercise time, change in Borg scale at rest vs. Borg scale at steady state vs. Borg at end exercise.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, double blind, crossover interventional design. The crossover allows for equality in number of subjects assigned to each treatment and for subjects to be their own controls. Baseline spirometry will be taken prior to exercise test. Subjects will be prepared for OEP. All exercise will take place on an electromagnetically braked cycle ergometer. Throughout the protocol heart rate, blood pressure, O2 saturation, ventilation, and metabolic data will be recorded. A modified exercise induced asthma protocol will be used. Unlike prior studies, ventilatory kinematics (with isolated diaphragmatic function) will be monitored throughout exercise using biomechanical motion analysis (OEP). This OEP analysis involves compartmentalization of the chest into three sections; 1) pulmonary rib cage, 2) diaphragmatic rib cage, and 3) abdomen to determine the contribution of each component to total lung volume. By measuring the percent contribution of compartment, we are able to better understand its impact on respiration. OEP will be able to quantify and assess the distortion effects of dynamic hyperinflation and obstruction.

Twenty moderate to severe COPD patients will be recruited. Subjects will refrain from their usual inhaled medications for 24 hours prior to the testing session. All subjects will be asked to verify that this is acceptable with their pulmonologist prior to participation. Subjects will also be asked to have their short acting bronchodilators and other regular medications available to be taken if symptoms should occur. During the initial screening, subjects will be familiarized with all procedures. Then baseline pulmonary function testing, and baseline resting OEP measurements will be performed. The subjects will then be randomized to receive either budesonide/formoterol fumarate dihydrate (Symbicort) or a placebo of budesonide only (Entocort EC). At that time, they will receive treatment with either placebo or budesonide/formoterol fumarate dihydrate and after 45 minutes, they will repeat spirometry and OEP and submaximal exercise testing with OEP. After one week, subjects will be tested again and switched to the opposite treatment (i.e. if on budesonide/formoterol fumarate dihydrate initially then switch to placebo and vice versa). The one week washout period between tests will include a resumption of the usual medications. The subjects will refrain from their inhaled medications for 24 hours before the second testing session, but use all of their other usual medications.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD by Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria
* Approval by pulmonologist
* Informed consent
* Age 40 to 75
* Males and females
* All races
* Ex smoker or non smoker
* Prior therapy allowed

Exclusion Criteria:

* No active cardiac disease
* Alpha1 Antitrypsin Deficiency
* Active smoking
* Reactive Airways Disease
* Pulmonary Hypertension
* Comorbid conditions preventing exercise (arthritic, neurologic, vascular, or other conditions)
* BMI>30
* Current enrollment in any other concurrent study at Columbia University Medical Center or sponsored by AstraZeneca at any other sites
* Participation in any pharmacologic studies in the last 6 months prior to enrollment in this study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bartels, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2013.
Groups:
- Active Medication or Placebo: Data per arm is not available. Columbia will never have access to this data.
Period: Overall Study
Arm/Group | Active Medication or Placebo
Started | 9
Completed | 8
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Medication or Placebo
Number analyzed (Participants) | 9
Age, Customized [Number; unit: participants]
  Between 40 and 75 years | 9
Sex/Gender, Customized [Number; unit: participants] — Gender breakdown is not available. Columbia will never have access to this data.
  participants
    Male and Female | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Change in Dynamic Hyperinflation Measured by End Expiratory Volumes Recorded by Optoelectronic Plethysmography (OEP).
Description: Our objective is to measure baseline, post treatment and post exercise spirometry and evaluate exercise dynamic hyperinflation before and after treatment using OEP. We hypothesize that budesonide/formoterol fumarate dihydrate will decrease dynamic hyperinflation as measured by OEP.
Time Frame: 2 hours
Population: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2013.
Arm/Group | Active Medication or Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Exercise Time in Steady State Exercise
Description: Our secondary objective is to evaluate duration of steady state exercise and exercise capacity before and after treatment. Our secondary hypothesis is that decreases in dynamic hyperinflation during exercise will lead to improvements in dyspnea with exercise, and allow for increases in exercise capacity.
Time Frame: 2 hours
Population: as for outcome 1
Arm/Group | Active Medication or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2013.
Arm/Group | Active Medication or Placebo
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No